CLINICAL TRIAL: NCT06626191
Title: Comparison of the Postoperative Analgesic Efficacy of Serratus Posterior Superior Intercostal Plane Block and Interscalene Brachial Plexus Block in Shoulder Arthroscopy
Brief Title: Comparison of the Postoperative Analgesic Efficacy of SPSIPB and ISBPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0073
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Arthroscopy; Peripheral Nerve Block; Pain Management
Keywords: Shoulder Arthroscopy; Interscalene Brachial Plexus Block; Serratus Posterior Superior Intercostal Plane Block
MeSH Terms: conditions — Agnosia | interventions — Population Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interscalene brachial plexus block (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, interscalene brachial plexus block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacaine) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Interscalene brachial plexus block
- Serratus posterior superior intercostal plane block (Active Comparator): After the patients are monitored and in the sitting position, after appropriate field sterilization, a serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacain) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Serratus posterior superior intercostal plane block
- Group without peripheral nerve block (Active Comparator): After the patients are monitored, they will be operated under general anesthesia without peripheral nerve block and intraoperative intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Group without peripheral nerve block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Interscalene brachial plexus block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacaine) under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Interscalene brachial plexus block
Procedure: Serratus posterior superior intercostal plane block — Patients will undergo serratus posterior superior intercostal plane block using 30 ml of local anesthetic solution (0.25% bupivacaine) under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Serratus posterior superior intercostal plane block
Procedure: Group without peripheral nerve block — In the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Group without peripheral nerve block

SUMMARY:
Shoulder arthroscopy is one of the common surgical procedures performed today. After shoulder surgery, providing adequate analgesia is necessary for both the comfort of the patient and the ability to perform the necessary post-operative rehabilitation exercises early and regularly.

Nerve blocks reduces opioid consumption in the postoperative period by providing better pain control and therefore has advantages such as fewer side effects and less risk of pulmonary and cardiac complications.

In this study; it was aimed to compare the analgesic effectiveness of interscalene brachial plexus block and serratus posterior superior intercostal plane block, with each other and with the control group in the postoperative period in patients who underwent shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II-III
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score IV and above
* Patients with a history of bleeding diathesis
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 24 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 0st, 1st, 2nd,4th, 12th, and 24th hours after surgery.

SECONDARY OUTCOMES:
Intraoperative remifentanil consumption Intraoperative opioid consumption | Intraoperative period
  Remifentanil consumption for intraoperative period will be recorded
Postoperative Tramadol Consumption | 24 hours after surgery
  Tramadol consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)